CLINICAL TRIAL: NCT04531592
Title: Evaluation of Valproic Acid (VPA) as Adjunctive Therapy for Liver Transplant Patients With Moderate to Severe Hemorrhage at Risk of Ischemia Reperfusion (I/R) Injury
Brief Title: Valproic Acid (VPA) for Acute Kidney Injury (AKI) in Liver Transplant Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by the Sponsor
Sponsor: Westat (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VPA-202
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury; Ischemia Reperfusion Injury
Keywords: valproic acid; acute kidney injury; ischemia reperfusion injury; hemorrhage; liver transplant
MeSH Terms: conditions — Acute Kidney Injury; Reperfusion Injury; Hemorrhage | interventions — Valproic Acid

STUDY DESIGN:
Intervention Model Description: A phase 2, single-dose, multicenter, double-blind, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: In addition to the individuals listed above, Sponsor's representatives such as clinical research associates who will perform site monitoring, the pharmacovigilance medical monitor, and all staff at the research sites other than the pharmacist of record will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VPA plus SOC (Experimental): A single dose of 140 mg/kg of VPA plus standard of care
  Interventions: Drug: Valproic acid
- Placebo plus SOC (Placebo Comparator): A single dose of isotonic saline solution plus standard of care
  Interventions: Drug: Isotonic saline solution

INTERVENTIONS:
Drug: Valproic acid — Valproate sodium in 5-ml single-dose vials containing 100 mg/ml of VPA. The appropriate dose of 140 mg/kg, based on the subject's weight at study entry, will be diluted in isotonic saline solution to a final volume of 300 ml for administration
  Other Names: valproate sodium
  Arms: VPA plus SOC
Drug: Isotonic saline solution — Isotonic saline solution consisting of 0.9% sodium chloride in the volume of 300 ml for administration
  Arms: Placebo plus SOC

SUMMARY:
The purpose of this study is to find out if a drug called valproic acid (VPA) will protect organs (like the kidneys) from harmful effects caused by the temporary drop and then rise of blood flow and oxygen (called ischemia reperfusion (I/R) injury that sometimes happens during liver transplant surgery. VPA is an approved drug for treating conditions such as seizures and migraines for many years. However, it is not approved for use at the higher dose that will be used in this study or for protecting organs from I/R injury. This study will enroll liver transplant patients and randomly assign them to receive either VPA diluted in salt water or salt water without VPA (placebo) and then follow the patients and compare their organ function and overall outcome. This study is masked meaning that the patients, doctors, and nurses will not know which patient received which treatment. The study treatment will be given in addition to the care that liver transplant patients normally receive. The researchers doing this study believe that VPA will lessen organ injury caused by I/R, meaning that patients who receive VPA will experience less kidney injury when compared to patients who receive the placebo.

DETAILED DESCRIPTION:
I/R injury remains a major clinical problem during liver transplantation. In addition to the implanted liver graft suffering from significant I/R injury due to the transplant process itself, other organs such as the kidneys frequently demonstrate significant I/R injury associated with substantial morbidity and mortality. Among liver transplant patients, especially those who have suffered significant blood loss and prolonged hypotension requiring multiple vasopressors, the rate of acute kidney injury (AKI) is reported to be >50%.

VPA is an anticonvulsant drug that was approved by the Food and Drug Administration (FDA) in 1978. VPA was developed for use as monotherapy or adjunctive therapy for the treatment of seizure disorders, mania associated with bipolar disorder, and migraine. Both oral and intravenous (IV) formulations are available. Doses up to 60 milligram (mg)/kilogram (kg)/day for up to 14 days have been demonstrated to be safe and effective. More recently, a study has shown that a single dose of intravenous VPA at up to 140 mg/kg is safe in healthy volunteers. VPA has been recognized as an HDAC inhibitor (HDACI) shown to reduce the inflammatory response and oxidative stress in septic mice, thereby protecting against renal injury. The molecular mechanisms conferring anticonvulsant properties associated with VPA have not been clearly elucidated to date but likely include increasing levels of γ-aminobutyric acid in the central nervous system (CNS), reduction in N-Methyl-D-Aspartate-mediated excitation, and blockade of voltage gated sodium and L-type calcium channels. More recently, VPA has shown HDACI potential, specifically targeting class I (subclasses Ia and Ib) and class II (subclass IIa) HDAC proteins. Given that VPA modulates multiple pathways involved in AKI, it theoretically could prevent kidney dysfunction and inflammation that is induced by I/R injury.

The aim of this study is to evaluate the effect of VPA on reducing I/R injury related to organ damage in the kidneys in liver transplant patients with moderate-to-severe hemorrhage. The primary objective is to evaluate the effect of VPA on reducing AKI compared with placebo in liver transplant patients with expected moderated-to-severe hemorrhage at risk for I/R injury. The two secondary objectives are: 1) To assess the perioperative pharmacokinetics (PK) of VPA in liver transplant patients with moderate-to-severe hemorrhage, and 2) To evaluate the safety of VPA administered as IV infusion in liver transplant patients with moderate-to-severe hemorrhage at risk of I/R injury.

This is a phase 2, single-dose, multicenter, double-blind, randomized, placebo-controlled study. Subjects will be randomized in a 1:1 ratio to receive a single dose of 140 mg/kg of VPA plus standard of care (SOC) or the placebo plus SOC, administered via IV infusion in the OR within 45 min after induction of anesthesia (administration of hypnotic). Clinical evaluations such as physical examination, vital signs, electrocardiogram, and laboratory results will be collected. AKI will be used to assess VPA efficacy. Myocardial injury and laboratory measurements (hematology, chemistry, coagulation profile, and urinalysis) will be used to monitor subject safety. Outcome measures including in-hospital mortality, length of intensive care unit (ICU) and/or stepdown unit (SDU) stay, length of hospital stay, number of alive and ventilator free days (aVFD), and incidence of renal replacement therapy (RRT) will also be collected. Blood samples will be collected for PK analysis. The PK analysis will correlate study drug exposures with safety profiles. Specimens (plasma, peripheral blood mononuclear cells (PBMCs), and urine) will be stored for future undetermined study-related analyses, including pharmacodynamics (PD) and VPA responsiveness studies. These studies may correlate PK profiles to molecular changes related to beneficial properties of VPA.

Male and non-pregnant, non-breastfeeding female liver transplant patients between 18 and 80 years old will be recruited for the study. Patients will be those scheduled to undergo liver transplant surgery and expected to require transfusion of 3 or more units of red cell product. Only patients who can provide consent or for whom a Legally Authorized Representative (LAR) can provide consent, will be enrolled. Approximately 50 subjects will be recruited from across four major medical centers for participation in this study.

Based on the available safety profile data from multi-dose clinical trials of VPA, the product safety information sheet, as well as the VPA Phase 1 study which evaluated the safety of single ascending doses of VPA, it has been determined that a dose of 140 mg/kg is safe and well-tolerated with minimal adverse reactions. However, given that patients studied at the 140 mg/kg dose in the phase 1 study were relatively healthy compared to the proposed patient population in this study and unanticipated Adverse Events (AEs) may occur, the study team will monitor all study subjects closely for AEs throughout the study. All AEs will be evaluated for duration, seriousness, severity, and relationship to the study drug, and reported accordingly.

This study will be monitored according to the data and safety monitoring plan which will outline the different levels of monitoring and the responsible parties. A Safety Review Committee (SRC) will review and monitor all safety information and compliance data as well as the overall study progress on a regular basis. A Medical Monitor (MM) with relevant clinical and research expertise will oversee the clinical study and provide ongoing medical monitoring. The clinical site Principal Investigators (PIs) will be responsible for ensuring that all AEs that occur in subjects during the AE reporting period are managed and reported in accordance with the protocol, Sponsor requirements, and any applicable regulations and institutional policies. A Data Monitoring Committee (DMC) will monitor implementation and progress of the study and review the accumulating endpoint and safety data by treatment arm to detect evidence of early significant benefit or harm for subjects while the study is in progress.

As the main purpose of this study is to evaluate safety of VPA in the study population and to investigate efficacy signal, this is a proof-of-concept (PoC) study. Because it is a PoC study rather than a confirmatory one, it has been assumed that a total sample size of 50 subjects (25 in each treatment arm) will be sufficient to provide adequate clinical evidence of safety and potential efficacy, and to support decision-making on whether a larger pivotal confirmatory Phase 3 study would be justified.

A statistical analysis plan (SAP) that details the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives will be developed. Demographic and relevant baseline characteristics will be presented and summarized descriptively by treatment for the randomized, modified intent-to-treat (mITT), and per-protocol (PP) populations. The primary endpoint of KDIGO stages will be measured in ordinal scale as 0, 1, 2, or 3, where 0 indicates normal renal function and the progressively higher values indicate worsening renal function. The ordinal scale measurements will be analyzed using the proportional odds ordinal logistic regression model. The KDIGO stages will be the dependent variable and drug treatment will be used as the independent variable. The common odds ratio across the KDIGO stages and its 95% confidence interval will be calculated. Binary endpoints (e.g., incidence of AKI) will be analyzed by Fisher's exact test or logistic regression with treatment as an independent variable. The odds ratio and its 95% confidence interval will be calculated. Continuous outcomes will be analyzed by missed effects models with treatment and baseline value of the outcome (if applicable) as independent variables. Un-ordered categorical variables with more than two levels of outcome will be analyzed by a chi-square test. Ordered categorical variables with more than two levels of outcome will be analyzed in the same way as for the primary endpoint. Safety endpoints will be analyzed and summarized descriptively. Categorical variables will be summarized by count and percentage. Odds ratios and relative risks may be calculated to compare study drug with placebo in incidence of certain safety events. Continuous variables will be summarized by mean, SD, median, minimum, and maximum. Shift tables may be used to describe changes in certain laboratory values. The plan for the PK analysis is two-fold. First, a standard noncompartmental analysis will be performed to obtain descriptors of VPA exposure to explore potential relationships to the primary outcome), secondary outcomes, or any observed adverse effects. A population PK analysis will be performed to examine and, perhaps, explain the anticipated differing PK of VPA in the trial. Specifically, low protein binding of VPA and massive blood loss are expected to affect the elimination clearance and, perhaps, the volume of distribution of VPA. Characterizing the degree to which the PK are perturbed as well as the parameter variability in this population will be important for analyzing the relationship of VPA exposure to primary and secondary outcomes and determining the effects, if any, of factors related to disease or perioperative conditions to the PK of VPA.

No interim analyses will be performed for this study. This study does not have a formal stopping rule based on statistical testing. See Section 3.9 for more information on stopping rules. Missing data can occur in clinical studies, and they may have an impact on the results of statistical analyses. Every effort will be made to ensure that the amount of missing data is kept at a minimum.

ELIGIBILITY:
Inclusion Criteria:

* Is aged 18 to 80 years old;
* Is male or non-pregnant, non-breastfeeding female;
* Is able to provide written informed consent or has an LAR from whom consent can be obtained;
* Body mass index (BMI) is between 18 kg/m2 and 35 kg/m2;
* Expected transfusion of 3 or more units of red cell product, as determined by the patient's provider; and
* Is scheduled to undergo liver transplant surgery without hepatocellular carcinoma (HCC) exception points.

Exclusion Criteria:

* Has a known history of adverse reaction to VPA;
* Is currently receiving VPA;
* Is pregnant or breastfeeding;
* Is in need of a simultaneous kidney transplant, or currently on RRT for either AKI or hepato-renal syndrome, type I (HRS-I);
* Is currently incarcerated or pending incarceration;
* Is known to have mitochondrial disorders caused by polymerase γ (POLG) mutations;
* Has acute liver failure;
* Has porto-pulmonary hypertension;
* Has hepato-pulmonary syndrome;
* Transplant procedure is a veno-venous bypass procedure;
* Is a living-donor transplant or a split liver transplant;
* Is scheduled to undergo liver transplant surgery with HCC exception points; or
* Has other unspecified reason/condition that, in the opinion of the clinical site PI, make the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Stage of AKI as assessed by Kidney Disease: Improving Global Outcomes (KDIGO) stage based on serum creatinine (SCr) | Within the first 48 hours after study drug administration
  The primary endpoint of AKI as assessed by KDIGO stages will be measured in ordinal scale as 0, 1, 2, or 3, where 0 indicates normal renal function and the progressively higher values indicate worsening renal function

SECONDARY OUTCOMES:
Blood lipocalin-2 (LCN2) | At baseline, 2 hours post reperfusion, 2 hours post ICU admission, and 24 hours post ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first
  LCN2 is an early biomarker of AKI
Urine lipocalin-2 (LCN2) | At baseline, 2 hours post reperfusion, 2 hours post ICU admission, and 24 hours post ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first
  LCN2 is an early biomarker of AKI
Incidence of AKI defined by the occurrence of KDIGO stages 1, 2, or 3 based on SCr, or based on urine output (UO) for those subjects with missing SCr | Within the first 48 hours after study drug administration
  Incidence of AKI defined by KDIGO stages where stage 0 is no occurrence of AKI and stages 1, 2, or 3 is occurrence of AKI. KDIGO staging will be based on SCr, or based on urine output (UO) for those subjects with missing SCr
Incidence of AKI defined by SCr increase or for those subjects with missing SCr, UO decrease | SCr upon ICU admission, at 12 hours, 24 hours, 36 hours, and 48 hours after ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first; or UO every 6 hours through 48 hours after study drug administration
  Incidence of AKI define by increase in SCr by ≥ 0.3 mg/ dl within 48 hours after study drug administration; or an increase in SCr to ≥ 1.5 times baseline anytime within the 7 days after study drug administration; or for those subjects with missing SCr, UO volume < 0.5 ml/kg/h for 6 hours
Estimated glomerular filtration rate (eGFR) based on SCr and/or cystatin C | Upon ICU admission, at 12 hours, 24 hours, 36 hours, and 48 hours after ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first
  eGFR to be calculated based on SCr and/or cystatin C using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

OTHER OUTCOMES:
Serum creatinine (SCr) values | Upon ICU admission, at 12 hours, 24 hours, 36 hours, and 48 hours after ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first
  Changes in SCr values through day of hospital discharge or Day 7 after study drug administration, whichever comes first
Volume of all fluids and blood products received by the subject | During and through 48 hours after study drug administration
  Volume of all fluids and blood products (including red blood cells (RBC), packed RBC, fresh frozen plasma, platelet, cryoprecipitate, and clotting factors) received by the subject
Timing of all fluids and blood products received by the subject | During and through 48 hours after study drug administration
  Timing of all fluids and blood products (including red blood cells (RBC), packed RBC, fresh frozen plasma, platelet, cryoprecipitate, and clotting factors) received by the subject
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | Daily through day of hospital discharge or Day 7, whichever comes first
  APACHE II score (minimum score = 0; maximum score = 71) as an assessment of disease severity. Higher score is associated with worst outcome
Intensive care unit (ICU) and/or stepdown unit (SDU) stay | Through Day 7 after study drug administration
  Length of time the subject remained in the ICU and/or SDU
Hospital stay | Through Day 7 after study drug administration
  Length of time the subject remained hospitalized
Renal replacement therapy (RRT) | Through Day 7 after study drug administration
  Incidence of RRT the subject required after study drug administration
Alive and ventilator free days (aVFD) | Through Day 7 after study drug administration
  Number of days that the subject was alive and ventilator free
Patient survival | Through Day 7 after study drug administration
  Whether or not subject is alive on Day 7 after study drug administration
Allograft survival | Through Day 7 after study drug administration
  Whether or not the allograft is alive on Day 7 after study drug administration
Myocardial injury | Upon ICU admission, at 12 hours, 24 hours, 36 hours, and 48 hours after ICU admission, and then daily through day of hospital discharge or Day 7, whichever comes first
  Number of subjects with myocardial injury defined by troponin I level greater than 0.04 nanogram/milliliter
Clavien-Dindo Classification | Daily through day of hospital discharge or Day 7, whichever comes first
  Clavien-Dindo classification (minimum grade = I; maximum grade = V) as a measure of surgical complication. Higher grade is associated with worst outcome
Treatment-emergent adverse events (TEAEs) | After study drug administration through Day 7
  Incidence of TEAEs
Adverse events of special interest (AESIs) | After study drug administration through Day 7
  Incidence of AESIs after a single infusion of VPA
Serious adverse events (SAEs) | After study drug administration through Day 7
  Incidence of SAEs
Deaths | After study drug administration through Day 7
  Incidence of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rabadan-Diehl, PharmD, PhD, Principal Investigator — Westat
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Denver, Denver, Colorado
  - University of Texas Southwest, Dallas, Texas
  - Houston Methodist Specialty and Transplant Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hilmi IA, Damian D, Al-Khafaji A, Planinsic R, Boucek C, Sakai T, Chang CC, Kellum JA. Acute kidney injury following orthotopic liver transplantation: incidence, risk factors, and effects on patient and graft outcomes. Br J Anaesth. 2015 Jun;114(6):919-26. doi: 10.1093/bja/aeu556. Epub 2015 Feb 10. PMID 25673576
- [Background] Georgoff PE, Nikolian VC, Bonham T, Pai MP, Tafatia C, Halaweish I, To K, Watcharotone K, Parameswaran A, Luo R, Sun D, Alam HB. Safety and Tolerability of Intravenous Valproic Acid in Healthy Subjects: A Phase I Dose-Escalation Trial. Clin Pharmacokinet. 2018 Feb;57(2):209-219. doi: 10.1007/s40262-017-0553-1. PMID 28497259
- [Background] Zheng Q, Liu W, Liu Z, Zhao H, Han X, Zhao M. Valproic acid protects septic mice from renal injury by reducing the inflammatory response. J Surg Res. 2014 Nov;192(1):163-9. doi: 10.1016/j.jss.2014.05.030. Epub 2014 May 20. PMID 24948542
- [Background] Chateauvieux S, Morceau F, Dicato M, Diederich M. Molecular and therapeutic potential and toxicity of valproic acid. J Biomed Biotechnol. 2010;2010:479364. doi: 10.1155/2010/479364. Epub 2010 Jul 29. PMID 20798865
- [Background] Li Y, Alam HB. Creating a pro-survival and anti-inflammatory phenotype by modulation of acetylation in models of hemorrhagic and septic shock. Adv Exp Med Biol. 2012;710:107-33. doi: 10.1007/978-1-4419-5638-5_11. PMID 22127890